CLINICAL TRIAL: NCT01710059
Title: Refined ADEPT: Human Augmentics for Sustained Wellbeing
Brief Title: Using Mobile Phones to Improve Adherence to Inhaled Steroids
Acronym: ADEPT4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Giselle Mosnaim, Principal Investigator, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 10010402; 5K23HL092292-04 (NIH)
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Asthma
Keywords: Health Status Disparities; Minority Health; Pediatrics; Behavioral Intervention; Cellular Phone; Peer Group
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental: Intervention Group (Experimental): Experimental: Intervention Group
  1) Asthma Supervision; 2) Mobile Phone with talking, texting, and data plan; 3) Inhaled Corticosteroid Mobile Phone Application to provide virtual doctor supervision, immediate feedback, and positive reinforcement for taking inhaled corticosteroid medication as indicated; and 4) Beta2-adrenergic agonist Mobile Phone Application to monitor real time patterns of use of beta2-adrenergic agonist medication for asthma.
  Interventions: Behavioral: Asthma Supervision; Behavioral: Mobile Phone; Behavioral: Inhaled Corticosteroid Mobile Phone Application; Behavioral: Beta2-adrenergic agonist Mobile Phone Application

INTERVENTIONS:
Behavioral: Asthma Supervision — Each participant will be provided with a spacer and a peak flow meter, and instructions on proper technique, by a member of the study team during the baseline period. They will also meet with study staff at study visits during the active treatment phase to review their adherence to daily inhaled corticosteroids and usage patterns of short acting B2-agonist medication.
Behavioral: Mobile Phone — Each participant will receive a mobile phone with talking, texting and a data plan. They will get to keep the mobile phone at the end of the study, but the talking, texting and data plan will only be active during their participation in the study.
Behavioral: Inhaled Corticosteroid Mobile Phone Application — The Inhaled Corticosteroid Mobile Phone Application will be used to provide virtual doctor supervision, immediate feedback, and positive reinforcement for taking inhaled corticosteroid medication as indicated.
Behavioral: Beta2-adrenergic agonist Mobile Phone Application — The Beta2-adrenergic agonist Mobile Phone Application will be used to track real time patterns of use of beta2-adrenergic agonist medication.

SUMMARY:
This study has two main goals. The first goal is to test whether a mobile phone intervention can increase adherence to daily inhaled steroid medications in African American adolescents prescribed this type of medication by his/her asthma doctor. The second goal is to use a mobile phone intervention to better understand real life patterns of use of quick-relief (beta2-adrenergic agonist) asthma medication in this population.

ELIGIBILITY:
Inclusion Criteria:

* 11-16 years of age
* self-identify as African American
* have persistent asthma
* be on a prescription daily inhaled corticosteroid medication for asthma
* be on a prescription inhaled beta2-adrenergic agonist medication for asthma

Exclusion Criteria:

* candidate refusal
* the presence of other co-morbidities that could interfere wtih study participation
* > 60% adherence to inhaled corticosteroid medication, measured by the electronic dose counter, during the run-in period

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Adherence to inhaled corticosteroids, measured objectively using an electronic dose counter | 10 weeks
  Adherence is measured as the mean of daily adherence to prescription inhaled corticosteroid dose over 14 days both at baseline and at week 10 of the active treatment phase. For the primary outcome, we will compare adherence at week 10 to adherence at baseline.

SECONDARY OUTCOMES:
To understand patterns of use of quick-relief medication for asthma | 10 weeks
  This study will use an electronic dose counter and mobile phone technology to track participants real time use of quick-relief (beta2-adrenergic agonist) medication for asthma during the 10 weeks of active treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle S. Mosnaim, MD, MS, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States